CLINICAL TRIAL: NCT01898299
Title: tDCS for Auditory Hallucinations in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Joshua Kantrowitz, Clinical Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6662
Record Dates: First submitted 2013-06-12; First posted 2013-07-12 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Direct Current Stimulation (Experimental): Transcranial Direct Current Stimulation (tDCS) treatments will take place for 20 minutes per day for 5 consecutive days
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): Sham tDCS(inactive)treatment (transcranial Direct Current Stimulation) will take place for 20 minutes per day for 5 consecutive days.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — A neurostimulation technique that passes an extremely weak electric current through the brain.
  Other Names: BrainStim SYS
  Arms: Transcranial Direct Current Stimulation
Device: Sham tDCS — Sham (inactive) tDCS treatment
  Arms: Sham tDCS

SUMMARY:
The purpose of the present research is to test a potential new treatment for auditory verbal hallucinations in schizophrenia that uses transcranial Direct Current Stimulation (tDCS), a neurostimulation technique that passes an extremely weak electric current through the brain. During the treatment, two electrodes are positioned on the scalp above regions of the brain implicated in abnormal cortical activity associated with auditory verbal hallucinations in schizophrenia. Due to the directional flow of current, one electrode, termed "cathodal",inhibits cortical activity, and the other, termed "anodal", increases cortical activity. These electrodes will be placed such that cathodal stimulation is applied to an area associated with hyperactivity and anodal stimulation to an area associated with hypoactivity. One preliminary study has revealed that this form of neurostimulation can alleviate auditory verbal hallucination symptoms both immediately following five days of treatment and up to three months after the final treatment. The goal of this study is to replicate these effects and explore the mechanisms that may underpin them.

DETAILED DESCRIPTION:
90 patients with persistent auditory verbal hallucinations will be recruited to this study. Each individual will participate in behavioral assessments lasting up to 3 hours each and will then be randomized to receive a series of active vs. sham tDCS treatments. For active treatment, patients will have the inhibitory (cathodal) tDCS electrode placed over left auditory cortex relative to an anodal placed over frontal cortex on the right side. tDCS treatments will take place for 20 min per day for 5 consecutive days. For sham, procedures will be similar except that sham (inactive) tDCS treatment will be used. Assessment batteries will then be repeated following completion of treatment and at 1 and 3 mo following treatment. In addition, patients will be offered the possibility to participate in a concurrent magnetic resonance imaging (MRI) study aimed at evaluating the effects of tDCS on activation of auditory cortex during an auditory discrimination task as well as on other imaging parameters related to resting brain activity and metabolism. Patients who agree to participate in this MRI study will be scanned before and after active or sham tDCS. In addition, 5-15 schizophrenia patients will complete a week of High-density, e.g., "high-definition" tDCS (HD-tDCS) open label.

In addition to hallucinating patients, we will recruit up to 20 healthy controls and 20 non-hallucinating patients, who will have similar assessments to the patients, but will not receive tDCS.

Overall, the investigators hypothesize that tDCS treatment will lead to reduction in hallucinations, improvement in auditory function, and change in EEG and MRI measurements so that patients more closely resemble healthy volunteers and non-hallucinating patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-55
* Structured Clinical Interview for DSM Disorders (SCID) primary diagnosis of DSM-IV (Diagnostic and Statistical Manual of Mental Disorders-Version IV) schizophrenia or schizoaffective disorder
* Persistent auditory verbal hallucinations
* Right handed
* Stable antipsychotic medication for > 4 weeks
* Normal hearing
* If female and not infertile, must agree to use one of the following forms of contraception for the duration of study participation: systemic hormonal treatment, an interuterine device (IUD) which was implanted at least 2 months prior to screening, or "double-barrier" contraception
* Willing/capacity to provide informed consent

Exclusion Criteria:

* Substance dependence or abuse (excluding nicotine) in the past 90 days
* Current significant laboratory abnormality
* History of seizure, epilepsy in self or fist degree relatives, stroke, brain surgery, head injury with loss of consciousness > 1 hour or clear cognitive sequelae, intracranial metal implants, known structural brain lesion, devices that may be affected by transcranial Direct Current Stimulation (tDCS) (pacemaker, medication pump, cochlear implant, implanted brain stimulator)
* Frequent and persistent migraines
* History of adverse reaction to neurostimulation or open skin wounds that would preclude safe placement of tDCS electrodes
* Participation in study of investigational medication/device within 4 weeks
* Current use of medications known to lower seizure threshold (lithium, serotonergic or tricyclic antidepressants)
* If female, pregnant or breast feeding at the time of screening
* For MRI study only: Claustrophobia or metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan, as determined according to the guidelines set forth in the following reference book: "Guide to MR procedures and metallic objects" Shellock, PhD, Lippincott-Raven press, NY 1998

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-07-14 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Javitt, MD, Principal Investigator — Nathan Kline Institute, New York State Psychiatric Institute
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - Nathan Kline Institute, Orangeburg, New York

REFERENCES:
- [Derived] Kantrowitz JT, Sehatpour P, Avissar M, Horga G, Gwak A, Hoptman MJ, Beggel O, Girgis RR, Vail B, Silipo G, Carlson M, Javitt DC. Significant improvement in treatment resistant auditory verbal hallucinations after 5 days of double-blind, randomized, sham controlled, fronto-temporal, transcranial direct current stimulation (tDCS): A replication/extension study. Brain Stimul. 2019 Jul-Aug;12(4):981-991. doi: 10.1016/j.brs.2019.03.003. Epub 2019 Mar 5. PMID 30922713

RESULTS

PARTICIPANT FLOW:
Period: Post Treatment (One Week)
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Started | 47 | 42
Completed | 47 | 42
Not Completed | 0 | 0
Period: Post Treatment (One Month)
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Started | 47 | 42
Completed | 44 | 38
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS | Total
Number analyzed (Participants) | 47 | 42 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (9.9) | 40.1 (8.6) | 39.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 32 | 35 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 40 | 34 | 74
  Unknown or Not Reported | 0 | 0 | 0
Auditory Hallucination Rating Scale (AHRS) total score [Mean (Standard Deviation); unit: units on a scale (total score)] — This is a seven item scale rating auditory hallucinations. Total score ranges from 1 to 41, with higher scores more severe.
  units on a scale (total score) | 24.8 (5.7) | 25.2 (5.7) | 25.0 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Severity of Refractory Auditory Hallucinations
Description: Total score: Auditory hallucinations as determined by Auditory Hallucinations Rating Scale (AHRS). This is a seven item scale rating auditory hallucinations. Total score ranges from 1 to 41, with higher scores more severe.
Time Frame: Auditory Hallucination Rating Scale score after one month
Population: Population at one month
Measure: Mean (Standard Deviation); unit: AHRS total score
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
Number analyzed (Participants) | 44 | 38
AHRS total score | 20.1 (9.9) | 23.1 (6.8)
Statistical Analysis 1: Comparison: Transcranial Direct Current Stimulation vs Sham tDCS; Test type: Superiority; p = 0.036, ANCOVA; Control for Chlopromazine equivalents; Cohen's d effectsize = 0.48

ADVERSE EVENTS:
Time Frame: 5 day treatment
Description: Adverse events >5%
Arm/Group | Transcranial Direct Current Stimulation | Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/42
Other Adverse Events (participants affected / at risk) | 0/47 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT01898299/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT01898299/SAP_001.pdf